CLINICAL TRIAL: NCT01529554
Title: Phase I-II Randomized Prospective Double-blind Multi-center Trial on the Effects of a Short Course of Oral Everolimus on Infarct Size, Left Ventricular Remodeling and Inflammation in Patients With Acute ST-Elevation Myocardial Infarction
Brief Title: Controlled Level EVERolimus in Acute Coronary Syndromes
Acronym: CLEVER-ACS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEVER-ACS
Record Dates: First submitted 2012-02-03; First posted 2012-02-09 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; ST-Elevation Myocardial Infarction; Infarct size; inflammation; everolimus
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Inflammation | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Active Comparator): Everolimus p.o. for 5 days (d0=7.5 mg, d1=7.5 mg, d2=7.5 mg, d3=5 mg, d4=5mg)
  Interventions: Drug: Everolimus
- Placebo (Placebo Comparator): Placebo comparator with identical composition of tablets except everolimus
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — (d0=7.5 mg, d1=7.5 mg. d2=7.5 mg, d3=5 mg, d4=5mg)
  Arms: Everolimus
Drug: Placebo — matched placebo tablets manufactured to be identical to verum tablets except content of everolimus
  Arms: Placebo

SUMMARY:
Acute myocardial infarction (AMI) constitutes the major cause of death in most nations and death rates and morbidity remain substantial in the years thereafter. Inflammation is a hallmark throughout the distinct stages of atherosclerotic lesion formation preceding AMI as well as at the time of plaque rupture and during the post-infarct repair phase. Harnessing its harmful consequences constitutes an attractive therapeutic approach to address this unmet medical need.

The objectives of this study are to evaluate the effects of mTOR inhibition (everolimus) on infarct size, myocardial function and inflammation in patients with ST-Elevation Myocardial Infarction.

The efficacy objectives are:

1. (1° endpoint):

   To assess the effect of mTOR inhibition (everolimus) on myocardial infarct size as change from baseline (12-72 hours after percutaneous coronary intervention) to 30 days follow-up measured by MRI (Late Gadolinium Enhancement (LGE) for transmurality).
2. (2° endpoint):

   To evaluate microvascular obstruction (MVO) as change from baseline (12-72 hours after percutaneous coronary intervention) to 30 days follow-up evaluated by MRI.
3. (3° endpoints):

   1. Change of left ventricular volume from baseline (12-72 hours after percutaneous coronary intervention) to 30 days follow-up measured by MRI.
   2. Change of biomarkers from time of coronary angiography to 30 days follow-up including a time-course (AUC). Biomarkers comprise hs-TnT, NT-proBNP, hs-CRP, IL-6 and inflammatory biomarkers OPG, sRANKL, OPN and CCN1.

The safety objectives are:

To explore the effect of mTOR inhibition (everolimus) on several clinical and safety laboratory parameters including plasma lipid levels and blood count. This will be complemented by analysis of inflammatory cell subsets in coronary thrombi and peripheral blood (CD4+ T helper lymphocyte subsets, monocyte subsets).

ELIGIBILITY:
Inclusion Criteria:

1. Elevation Myocardial Infarction (STEMI) as defined by:

   * ST-Elevation > 1mm in > 2 leads OR
   * Novel left bundle branch block (LBBB) OR
   * Posterior MI with ST-Depression > 1mm in > 2 leads
2. Chest pain duration of > 10 minutes
3. Primary Coronary Intervention (PCI) with drug-eluting stent (DES) within 24 hours of chest pain onset in the occluded culprit artery
4. First Myocardial Infarction
5. Occluded coronary artery at angiography specifically occlusion of one coronary vessel in the proximal third of either LAD, RCX or RCA, the mid segment of right coronary artery (RCA) or mid segment of a large left anterior descending (LAD) coronary artery, i.e. when the latter reaches the apex.
6. Male and female patients 18 years to 90 years of age
7. Signed informed consent

Exclusion Criteria:

1. Participation in another drug or stent trial
2. Pregnant women or nursing mothers
3. Mechanical complication during acute coronary syndrome
4. Scheduled PCI for additional lesion within 30 days
5. Multivessel disease
6. Major elective surgery planned in trial period
7. Malignancy (unless healed or remission > 5 years)
8. Chronic infection (HIV, Tbc, empyema)
9. Severely compromised renal function (GFR< 30 ml/min)
10. Positive PCR Test for SARS-CoV-2 and/or at least one positive answer to questions regarding symptoms/contact related to COVID-19.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size measured by MRI | Change from baseline at 30 days
  To assess the effect of mTOR inhibition (everolimus) on myocardial infarct size as measured by MRI (Late Gadolinium Enhancement (LGE) for infarct size (transmurality) at 12-72 h (baseline) and 30 days

SECONDARY OUTCOMES:
Microvascular obstruction (MVO) measured by MRI | Change from baseline at 30 days
  To evaluate microvascular obstruction (MVO) by MRI at 12-72 h (baseline) and 30 days

OTHER OUTCOMES:
Left ventricular volume measured by MRI | Change from baseline at 30 days
  To evaluate left ventricular volume by MRI at 12-72 h (baseline) and 30 days
Biomarkers | Change from baseline at 30 days including time course
  To evaluate the changes of left ventricular volume from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, Professor, Study Director — UniversityHospitalZurich
Locations (8):
- Germany (4):
  - Kerckhoff-Klinik, Department of Cardiology, Bad Nauheim
  - University Hospital Chartié, Berlin
  - University Hospital Duesseldorf, Düsseldorf
  - University Hospital Mainz, Mainz
- Switzerland (4):
  - University Hospital Bern, Bern
  - University Hospital Geneva, Geneva
  - Cardiocentro Ticino, Lugano
  - University Hospital Zurich, Zurich

REFERENCES:
- [Derived] Candreva A, Gotschy A MD PhD, Stehli J, Bissig L, Lodi Rizzini M, Chiastra C, Gallo D, Morbiducci U, Klingenberg R, Heg D, Matter CM, Ruschitzka F, Manka R, Stahli BE. Microcirculatory Resistance After Primary Percutaneous Coronary Intervention Predicts Residual Myocardial Damage and Scar Formation. J Am Heart Assoc. 2025 Feb 18;14(4):e036033. doi: 10.1161/JAHA.124.036033. Epub 2025 Feb 8. PMID 39921502
- [Derived] Stahli BE, Klingenberg R, Heg D, Branca M, Manka R, Kapos I, Muggler O, Denegri A, Kesterke R, Berger F, Stehli J, Candreva A, von Eckardstein A, Carballo D, Hamm C, Landmesser U, Mach F, Moccetti T, Jung C, Kelm M, Munzel T, Pedrazzini G, Raber L, Windecker S, Templin C, Matter CM, Luscher TF, Ruschitzka F. Mammalian Target of Rapamycin Inhibition in Patients With ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2022 Nov 8;80(19):1802-1814. doi: 10.1016/j.jacc.2022.08.747. Epub 2022 Aug 29. PMID 36049557
- [Derived] Klingenberg R, Stahli BE, Heg D, Denegri A, Manka R, Kapos I, von Eckardstein A, Carballo D, Hamm CW, Vietheer J, Rolf A, Landmesser U, Mach F, Moccetti T, Jung C, Kelm M, Munzel T, Pedrazzini G, Raber L, Windecker S, Matter CM, Ruschitzka F, Luscher TF. Controlled-Level EVERolimus in Acute Coronary Syndrome (CLEVER-ACS) - A phase II, randomized, double-blind, multi-center, placebo-controlled trial. Am Heart J. 2022 May;247:33-41. doi: 10.1016/j.ahj.2022.01.010. Epub 2022 Jan 28. PMID 35092722